CLINICAL TRIAL: NCT00594126
Title: A Phase 1 Sequential Cohort, Dose Escalation Trial to Determine the Safety, Tolerability, and Maximum Tolerated Dose of GRN163L in Patients With Refractory or Relapsed Multiple Myeloma
Brief Title: Safety and Dose Study of GRN163L Administered to Treat Patients With Refractory or Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Geron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP14A004
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Multiple Myeloma; Relapsed Multiple Myeloma; Refractory Multiple Myeloma; Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Recurrence | interventions — imetelstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): 3+3 cohort dose escalation
  Interventions: Drug: Imetelstat Sodium (GRN163L)

INTERVENTIONS:
Drug: Imetelstat Sodium (GRN163L) — 25% dose escalation infused over 2 hours weekly

SUMMARY:
The purpose of this study is to determine the safety and the maximum tolerated dose (MTD) of GRN163L when administered to patients with refractory or relapsed multiple myeloma.

DETAILED DESCRIPTION:
GRN163L is a telomerase template antagonist with in vitro and in vivo activity in a variety of tumor model systems. Telomerase is an enzyme that is active primarily in tumor cells and is crucial for the indefinite growth of tumor cells. Inhibition of telomerase may result in antineoplastic effects.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple myeloma (either secretory or nonsecretory disease)
* Relapsed or refractory disease
* At least two prior treatment regimens
* ECOG performance status 0-2
* Adequate hepatic/renal function and platelet count
* If previously treated with an anthracycline, anthracenedione, or trastuzumab, must have left ventricular ejection fraction > 50%

Exclusion Criteria:

* Prior allogeneic bone marrow transplant, including syngeneic transplant
* Known intracranial disease or epidural disease
* Prior malignancy (within the last 3 years)
* Clinically significant cardiovascular disease or condition
* Active or chronically recurrent bleeding (eg, active peptic ulcer disease
* Prolongation of PT or aPTT > the ULN or fibrinogen < the LLN
* Clinically relevant active infection
* Serious co-morbid medical conditions, including cirrhosis and chronic obstructive or chronic restrictive pulmonary disease
* Symptomatic hyperviscosity syndrome
* Any other cancer therapy within 3 weeks prior to study, except for mitomycin C, nitrosoureas, or high-dose chemotherapy with stem cell support within 6 weeks prior to study
* Investigational therapy within 4 weeks prior to study
* Anti-platelet therapy within 2 weeks prior to study, other than low dose aspirin prophylaxis therapy and low dose heparin administration for management of IV access devices
* Radiation therapy within 4 weeks prior to study
* Major surgery within 4 weeks prior to study
* Active autoimmune disease requiring immunosuppressive therapy
* Known positive serology for HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Safety and MTD | First 3 weeks

SECONDARY OUTCOMES:
PK, PD, and efficacy | Baseline to end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Steve Kelsey, MD, Study Director — Geron Corporation
Locations (3):
- United States (3):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins University, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York

REFERENCES:
- See also: Related Info — http://www.geron.com